CLINICAL TRIAL: NCT06693388
Title: Whole-body Vibration for Children with Cerebral Palsy Undergoing Serial Casting
Brief Title: WBV and Serial Casting for Children with Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ben Reader (Other)
Responsible Party: Sponsor-Investigator, Ben Reader, Research Scientist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00004078
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy (CP); Cerebral Palsy
Keywords: Serial Casting; Whole body Vibration; Cerebral Palsy; Pediatrics
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Serial Casting Only (Active Comparator)
  Interventions: Other: Serial Casting
- Serial Casting + Exercise (Active Comparator)
  Interventions: Other: Exercise; Other: Serial Casting
- Serial Casting + Exercise + WBV (Active Comparator)
  Interventions: Other: Exercise; Other: Whole-Body Vibration; Other: Serial Casting

INTERVENTIONS:
Other: Exercise — 2 minutes each exercise with 30 sec break - 4 exercises prior to serial casting
  Arms: Serial Casting + Exercise; Serial Casting + Exercise + WBV
Other: Whole-Body Vibration — WBV prior to serial casting
  Arms: Serial Casting + Exercise + WBV
Other: Serial Casting — Serial Casting as provided by standard of care

SUMMARY:
Children with cerebral palsy have increased muscle tone which often results in decreased active and passive movement at the ankle. While many management strategies exist (including passive stretching, WBV, serial casting, Botox, and surgical tendon lengthening), the utilization of WBV in combination with active exercises and serial casting has not been previously explored. Serial casting is the repeated application of a fiberglass cast (such as that applied to manage stable fractures) on a scheduled (usually weekly basis) to gradually increase the range of motion at a specific joint. It is theorized that combining previously established standard of care practices may result in more rapid clinical change, and hence reduce the need for prolonged intervention; ultimately reducing healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-17 and 32 weeks exclusive years;
* Diagnosis of cerebral palsy;
* GMFCS levels I-III;
* Stands with upper extremity support or less support;
* Active referral from a prescribing provider for serial casting with ankle DF of <10 degrees;
* Willing to pursue care at [primary site] outpatient physical therapy clinic for the duration of the study;
* Subjects/families must be able to communicate in the English language without the need for interpreter.

Exclusion Criteria:

* History of selective dorsal rhizotomy;
* previous Achilles tendon lengthening or other orthopedic interventions to the lower extremities in 1 year prior to enrollment;
* No Botox or changes in oral medication to reduce spasticity within 6 months prior to enrollment;
* skin, circulation, vascular conditions;
* Previous history of cancer;
* Reduced ankle/foot sensation;
* Allergies to casting materials.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ankle Dorsiflexion Range of Motion (Goniometer) | Longitudinal through study completion, an average of 6 weeks but upto 12 weeks
  Measured with Goniometer in degrees. Knee flexed and knee extended.

SECONDARY OUTCOMES:
Pain (Visual Analogue Scale/Wong-Baker Faces) | Longitudinal through study completion, an average of 6 weeks but upto 12 weeks
  Wong-Baker Faces will be used for those unable to provide a visual analogue scale score. Visual Analogue Scale = 0 (no pain) - 10 (worst pain). Wong-Baker Faces = ordinal level categories of pain. Categories = 0 no hurt, 2 hurts little bit, 4 hurts little more, 6 hurts even more, 8 hurst whole lot, 10 hurts worst. On both scales, higher number will be worst outcomes.
Length of Casting Episode (Weeks) | Longitudinal through study completion, an average of 6 weeks but upto 12 weeks
  Measured in weeks from the date of first serial cast application to date of last cast applied. This will be extracted from the electronic health record.

OTHER OUTCOMES:
Adverse effects | Longitudinal through study completion, an average of 6 weeks but upto 12 weeks
  skin breakdown, early removal etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No